CLINICAL TRIAL: NCT04535284
Title: Coaching Intervention for Caregivers of Persons With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20D.718
Record Dates: First submitted 2020-08-06; First posted 2020-09-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Caregiver Stress Syndrome; Caregiver Burnout; Stroke, Acute
Keywords: Caregiver; Stroke; Coaching; Stress; Self-efficacy; Re-admission; Burden
MeSH Terms: conditions — Caregiver Burden; Stroke

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial design with two parallel groups
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded to treatment group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching (Experimental): Health Coaching-in-Context" includes coaching by trained coaches up to 10 sessions over teleconference.
  Interventions: Behavioral: Coaching
- Usual Care (No Intervention): The usual care group does not get any intervention but continues with any of their usual activities that would otherwise would have been provided to them.

INTERVENTIONS:
Behavioral: Coaching — "Health Coaching-in-Context" that consists of up to 10 sessions, arranged once-a-week or multiple times a week based on convenience of scheduling for up to 10 weeks. The program targets improved caregiver health through occupational therapy coaching.
  Other Names: Health Coaching in Context
  Arms: Coaching

SUMMARY:
Caregivers of people with stroke experience strain that can reduce their quality of life. Caregivers are routinely engaged during hospital discharge for education and training related to the person with stroke. However, the critical period after stroke survivor's discharge is largely unsupported for the caregiver. This proposed study is a randomized controlled trial that will provide post-discharge support for caregivers using a health coaching program as compared to usual care and examine its effect of caregivers and people with stroke.

DETAILED DESCRIPTION:
Caregiver strain reduces quality of life and can increase the chance of unplanned hospital readmission for the person with stroke. Caregivers are routinely engaged during hospital discharge for education and training. However, the critical period after discharge is largely unsupported. The proposed research will integrate occupational therapy and telehealth to provide a post-discharge, caregiver-focused program, the "Health Coaching-in-Context" that consists of up to 10 sessions, arranged once-a-week or multiple times a week based on convenience of scheduling for up to 10 weeks. The program targets improved caregiver health and reduction in readmissions for stroke survivor. The study aims to examine the effects of the coaching program for caregivers as compared to usual care and evaluate the feasibility of study design. A pilot randomized controlled trial will be conducted with two parallel groups, "Health Coaching-in-Context" and usual care. A sample of up to 40 pairs, including up to 40 stroke survivors and their respective 40 caregivers will be recruited from University hospitals and randomly assigned after consenting. The occupational therapist, unaware of the group assignment, will administer assessments before and after the intervention, and at 4-week follow-up. Data will be collected on general information, readmissions, performance, self-efficacy, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Survivor criteria: First-time stroke, discharged from hospital within the past 30 days.
* Caregiver criteria: Informal caregiver primarily responsible for care (family member, friend, or partner), may or may not live in the same household. Passes cognition screen, willing to use teleconference using phone, tablet, or computer.
* Both: 18 to 80 years of age, understand and speak English

Exclusion Criteria:

* Children
* 81 years of age or older
* Unable to understand and speak English
* Does not provide consent
* Caregiver does not pass cognition screen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Week 1
  Measure of performance and satisfaction with performance of daily tasks. Each domain score is out of 10, minimum is 1, and higher scores are better.
Canadian Occupational Performance Measure | Week 12
  Measure of performance and satisfaction with performance of daily tasks.Each domain score is out of 10, minimum is 1, and higher scores are better.
Canadian Occupational Performance Measure | Week 15
  Measure of performance and satisfaction with performance of daily tasks. Each domain score is out of 10, minimum is 1, and higher scores are better.

SECONDARY OUTCOMES:
Re-admission | 30 day re-admission
  Number of subjects readmitted. Lower is better.
Re-admission | 60 day re-admission
  Number of subjects readmitted. Lower is better.
Re-admission | 90 day re-admission
  Number of subjects readmitted. Lower is better.
Revised Caregiver Self-efficacy scale | Week 1
  Measure of confidence with caregiving related tasks. 0 to 100 range for 15 items, higher score is better self-efficacy
Revised Caregiver Self-efficacy scale | Week 12
  Measure of confidence with caregiving related tasks. 0 to 100 range for 15 items, higher score is better self-efficacy
Revised Caregiver Self-efficacy scale | Week 15
  Measure of confidence with caregiving related tasks. 0 to 100 range for 15 items, higher score is better self-efficacy
Zarit Burden Interview | Week 1
  Burden experienced by caregiver while caring for person with stroke. Lower score is better, 22 items, range is 0 to 88.
Zarit Burden Interview | Week 12
  Burden experienced by caregiver while caring for person with stroke. Lower score is better, 22 items, range is 0 to 88.
Zarit Burden Interview | Week 15
  Burden experienced by caregiver while caring for person with stroke. Lower score is better, 22 items, range is 0 to 88.
WHO-BREF Quality of Life scale | Week 1
  World Health Organization-Brief Quality of life evaluation. Higher Scores are better. Scores in four domains 0 to 100 each
WHO-BREF Quality of Life scale | Week 12
  World Health Organization-Brief Quality of life evaluation. Higher Scores are better. Scores in four domains 0 to 100 each
WHO-BREF Quality of Life scale | Week 15
  World Health Organization-Brief Quality of life evaluation. Higher Scores are better. Scores in four domains 0 to 100 each
Single-item life satisfaction scale | Week 1
  Life Satisfaction Evaluation. Lower scores are better, range from 1 to 4 Satisfaction with life - one question Quality of life evaluation Satisfaction with life - one question Quality of life evaluation Satisfaction with life - one question Satisfaction with life - one question
Single-item life satisfaction scale | Week 12
  Life Satisfaction Evaluation. Lower scores are better, range from 1 to 4 Satisfaction with life - one question Quality of life evaluation Satisfaction with life - one question Quality of life evaluation Satisfaction with life - one question Satisfaction with life - one question
Single-item life satisfaction scale | Week 15
  Life Satisfaction Evaluation. Lower scores are better, range from 1 to 4 Satisfaction with life - one question Quality of life evaluation Satisfaction with life - one question Quality of life evaluation Satisfaction with life - one question Satisfaction with life - one question
Stroke Impact Scale | Week 1
  The impact of stroke on various areas of daily activities of the person with stroke. Range from 0 to 100, higher is better.
Stroke Impact Scale | Week 12
  The impact of stroke on various areas of daily activities of the person with stroke. Range from 0 to 100, higher is better.
Stroke Impact Scale | Week 15
  The impact of stroke on various areas of daily activities of the person with stroke. Range from 0 to 100, higher is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared within the research team. De-identified data will be made publicly available on a repository.